CLINICAL TRIAL: NCT04578028
Title: A Randomised, Double Blind, Placebo Controlled, Single Centre, Three-Part Study to Assess the Safety, Tolerability and Pharmacokinetics of Single and Multiple Oral Doses of ONO-2808 in Healthy Subjects.
Brief Title: A First in Human Study to Assess the Safety, Tolerability and Pharmacokinetics of ONO-2808-01 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ono Pharmaceutical Co. Ltd (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: ONO-2808-01; 2019-004693-26 (EudraCT Number)
Record Dates: First submitted 2020-10-01; First posted 2020-10-08 (Actual); Last update posted 2021-12-30 (Actual); Status verified 2021-12

CONDITIONS: Neurodegenerative Diseases
Keywords: Neurodegenerative Diseases
MeSH Terms: conditions — Neurodegenerative Diseases

STUDY DESIGN:
Intervention Model Description: This is a single centre, three-part study conducted at a specialised Phase I centre to evaluate the safety, tolerability and pharmacokinetics of ONO-2808. This study consists of: Part A single ascending dose (including an assessment of potential food effects), Part B an assessment of age, and Part C multiple ascending dose. All parts of the study are conducted in healthy male and female (women of non-child bearing potential) participants. All parts of the study will have a 28-day screening period followed by admission to the clinical unit at least one day prior to dosing (Day -1) for baseline assessments. For all Parts of the study, a sentinel dosing approach is used to mitigate the overall safety risk with at least 1 day stagger to the rest of the cohort.
Who Masked: Participant, Investigator
Masking Description: This is a double-blind study. A sentinel dosing approach will be used in the study at each new ascending dose level in Part A, B, and C. To maintain the blinded nature of the study, the sentinel participants will be randomised to drug or placebo in a 1:1 ratio.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- ONO-2808 Part A - Fasted (Experimental): Single ascending doses of ONO-2808 or placebo orally under fasted conditions. Additional descriptive information (including which interventions are administered in each arm) to differentiate each arm from other arms in the clinical trial.
  Interventions: Drug: ONO-2808
- ONO-2808 Placebo Part A- Fasted (Placebo Comparator): Single ascending doses of ONO-2808 or placebo orally under fasted conditions
  Interventions: Drug: Placebo
- ONO-2808 Part A - Fed (Experimental): Single ascending doses of ONO-2808 or placebo orally under fed conditions
  Interventions: Drug: ONO-2808
- ONO-2808 Placebo Part A - Fed (Placebo Comparator): Single ascending doses of ONO-2808 or placebo orally under fed conditions
  Interventions: Drug: Placebo
- ONO-2808 Part B (Experimental): Single dose of ONO-2808 or placebo in elderly female or elderly male healthy volunteers .
  Interventions: Drug: ONO-2808
- ONO-2808 Placebo Part B (Placebo Comparator): Single dose of ONO-2808 or placebo in elderly female or elderly male healthy volunteers
  Interventions: Drug: Placebo
- ONO-2808 Part C (Experimental): Multiple ascending doses of ONO-2808 or placebo orally
  Interventions: Drug: ONO-2808
- ONO-2808 Placebo Part C (Placebo Comparator): Multiple ascending doses of ONO-2808 or placebo orally
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ONO-2808 — Investigational drug
  Arms: ONO-2808 Part A - Fasted; ONO-2808 Part A - Fed; ONO-2808 Part B; ONO-2808 Part C
Drug: Placebo — Placebo drug
  Arms: ONO-2808 Placebo Part A - Fed; ONO-2808 Placebo Part A- Fasted; ONO-2808 Placebo Part B; ONO-2808 Placebo Part C

SUMMARY:
This is a first in human study to determine the safety, tolerability and pharmacokinetics of ONO-2808 in healthy adult participants. The study will be conducted in 3 parts: Part A, a single-ascending dose part with an assessment of the potential food effects in non-Japanese adult participants; Part B, a single dose part to assess the effect of age in non-Japanese elderly participants; and Part C, a multiple-ascending dose part with ONO-2808 administered to healthy subjects.

ELIGIBILITY:
Inclusion criteria:

1. Able to provide fully informed written consent.
2. 18-55 years (Part A & C) or ≥65 years (Part B).
3. Male and female participants (Women of non-child bearing potential (WONCBP)).
4. Agree to use an effective method of contraception.
5. No clinically significant medical history and no abnormal physical examination, laboratory profiles, vital signs or ECG abnormalities, based on the Screening examination.
6. Body mass index (BMI) of ≥18.5 to <30 kg/m2 and a body weight of at least 50 kg for males and 45 kg for females to a maximum of 100 kg, at the time of screening.
7. Estimated Creatinine Clearance (CrCL, Cockcroft-Gault equation) ≥90 mL/min at Screening. In Part B only, an estimated CrCL of ≥60mL/min at Screening.

Exclusion Criteria:

1. Mentally or legally incapacitated or with significant emotional problems at the time of the Screening visit or expected during the conduct of the study.
2. History or presence of clinically significant medical, surgical or psychiatric condition (including history of suicidal behaviour) or objection by General Practitioner (GP) to participant entering trial.
3. Liver chemistry values above the upper limit of normal (ULN) at Screening or admission.
4. Sensitivity to the study drug.
5. Female who is pregnant or lactating or of childbearing potential.
6. History or presence of alcoholism or drug/chemical/substance abuse.
7. Evidence of poor venous access as assessed by PI.
8. Use of any medication which may affect ONO-2808 pharmacokinetics or pharmacodynamics
9. Current smoker or has smoked (including use of tobacco and/or nicotine-containing products) in the previous 3 months
10. Positive urine drugs of abuse, cotinine or alcohol results at Screening or admission.
11. Positive results for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg) or hepatitis C virus (HCV).
12. Supine resting blood pressure less than 90/40 millimeter of mercury (mmHg) or greater than 140/90 mmHg (Part A& C) and less than 90/40 mmHg or greater than 160/90 mmHg (Part B).
13. Supine resting pulse rate lower than 40 beats per minute (bpm) or higher than 100 bpm.
14. Clinically significant history or presence of ECG findings at screening.
15. Use of any drug, including prescription and non-prescription medications, herbal remedies, or vitamin supplements within 14 days or five half-lives (whichever is longer) of first dosing and throughout the study.
16. Consumption or intake of compounds, food or fluids that are known to be a substrate, inducer or inhibitor of CYP450 for 28 days prior to the first dosing and throughout the study.
17. Donation of blood or significant blood loss within 56 days prior to the first dosing, or plasma donation within 7 days prior to the first dosing.
18. Participation in another clinical study within the last 3 months (or 5 half-lives of the study drug, whichever is longer) prior to the first dosing.
19. Objection by PI
20. Participants who are not willing to eat a high fat breakfast

    Exclusion criteria, applicable to all participants undergoing lumbar puncture for CSF collection (Part A & C):
21. History of significant back pain, significant kyphosis and or scoliosis or other spinal column deformities.
22. History or evidence of fundoscopy suggestive of raised intracranial pressure.
23. History or presence of any allergy or contraindication to the local anaesthetic required for participants undergoing lumbar puncture.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2020-08-19 (Actual); Primary Completion 2021-08-26 (Actual); Study Completion 2021-10-07 (Actual)

PRIMARY OUTCOMES:
Treatment emergent adverse events (TEAEs) by severity. | Part A and B: up to day 7; Part C: up to 17 days.
  Number of participants with TEAEs. An adverse event is any untoward medical occurrence in a participant who receive study drug without regard to possible causal relationship.
Serious adverse events (SAEs) | Part A and B: up to day 7; Part C: up to 17 days.
  Number of participants with SAEs. An SAE is an AE resulting in any of the following outcomes or deemed significant for any other reason: death, initial or prolonged hospitalization, life-threatening experience or persistent disability.
Vital signs | Part A and B: up to day 7; Part C: up to 17 days
  Summary statistics of vital signs and number of participants with clinically significant changes in vital signs including pulse/heart rate, respiratory rate, and blood pressure
ECG parameters | Part A and B: up to day 7; Part C: up to 17 days.
  Number of participants with ECG abnormalities
Clinical laboratory tests | Part A and B: up to day 7; Part C: up to 17 days
  Number of participants with clinical laboratory abnormalities (including haematology, clinical chemistry and urinalysis)
Physical examination | Part A and B: up to day 7; Part C: up to 17 days
  Number of participants with physical examination abnormalities
Neurological examination | Part A and B: up to day 7; Part C: up to 17 days.
  Number of participants with neurological examination abnormalities
Number of participants with suicidal behaviour | Part C: up to 17 days
  Treatment-emergent suicidal ideation and behaviour will be monitored by using the Columbia Suicide Severity Rating Scale (C-SSRS) and reported.

SECONDARY OUTCOMES:
Pharmacokinetics (Cmax) | Part A & B: Day 1 through Day 7, Part C: Day 1 and 14
  Assessment of the maximum observed plasma concentration of ONO-2808
Pharmacokinetics (Tmax) | Part A & B: Day 1 through Day 7, Part C: Day 1 and 14
  Assessment of the time to reach Tmax for ONO-2808
Pharmacokinetics (AUClast) | Part A & B: Day 1 through Day 7
  Assessment of the area under the concentration-time curve of ONO-2808 to last measurable concentration
Pharmacokinetics (AUCinf) | Part A & B: Day 1 through Day 7
  Assessment of the area under the concentration-time curve of ONO-2808 extrapolated to infinite time in plasma
Pharmacokinetics (AUCtau) | Part C: Day 1 and Day 14
  Assessment of the area under the concentration-time curve of ONO-2808 during the dosing interval in plasma
Pharmacokinetics (T1/2) | Part A & B: Day 1 through Day 7
  Assessment of the terminal elimination half-time of ONO-2808 in plasma
Pharmacokinetics (CL/F) | Part A & B: Day 1 through Day 7
  Assessment of the apparent clearance of ONO-2808 from plasma
Pharmacokinetics (Vz/F) | Part A & B: Day 1 through Day 7
  Assessment of the apparent volume of distribution of ONO-2808 during terminal elimination phase
Pharmacokinetics (Aetz) | Part A & B: Day 1 through Day 5, Part C: Day 1, 8 & 14
  Assessment of the amount of ONO-2808 excreted in urine over the period of sample collection
Pharmacokinetics (Percentage fe) | Part A & B: Day 1 through Day 5, Part C: Day 1, 8 & 14
  Assessment of the cumulative percentage of orally administered ONO-2808 excreted into urine
Pharmacokinetics (CLR) | Part A & B: Day 1 through Day 5, Part C: Day 1, 8 & 14.
  Assessment of the renal clearance of ONO-2808 from plasma
Distribution of ONO-2808 to the brain in Part A | Part A (in selected fasted cohorts): Day 1 and 2, Part C: Day 1 and Day 14
  Assessment of ONO-2808 brain distribution by measuring drug concentration in the cerebro spinal fluid (CSF)

CONTACTS AND LOCATIONS:
Overall Officials: Pablo F Soto, MD,MSc, PhD, Principal Investigator — Parexel
Locations (1):
- Parexel International Early Phase Clinical Unit (EPCU), London, United Kingdom

IPD SHARING:
Plan to Share IPD: No